CLINICAL TRIAL: NCT03677934
Title: Phase III, Multicenter, Randomized, Visual Assessor-Masked, Active-Comparator Study of the Efficacy, Safety, and Pharmacokinetics of the Port Delivery System With Ranibizumab in Patients With Neovascular Age-Related Macular Degeneration
Brief Title: A Phase III Study to Evaluate the Port Delivery System With Ranibizumab Compared With Monthly Ranibizumab Injections in Participants With Wet Age-Related Macular Degeneration
Acronym: Archway
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GR40548
Record Dates: First submitted 2018-09-11; First posted 2018-09-19 (Actual); Results first posted 2022-03-25 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-09

CONDITIONS: Neovascular Age-Related Macular Degeneration
MeSH Terms: interventions — Ranibizumab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PDS Implant Arm (Experimental): Participants will receive ranibizumab delivered through the PDS implant with 100 mg/mL in the study eye on Day 1 and receive refill-exchanges at fixed 24-week intervals
  Interventions: Drug: PDS Implant filled with 100 mg/mL Ranibizumab
- Intravitreal Arm (Active Comparator): Participants will receive ranibizumab 0.5 mg monthly intravitreal injections of 10 mg/mL formulation at Day 1 and every month thereafter.
  Interventions: Drug: Intravitreal Injections of 10 mg/mL Ranibizumab

INTERVENTIONS:
Drug: PDS Implant filled with 100 mg/mL Ranibizumab — Will be administered as per the schedule described in individual arm.
  Arms: PDS Implant Arm
Drug: Intravitreal Injections of 10 mg/mL Ranibizumab — Will be administered as per the schedule described in individual arm.
  Arms: Intravitreal Arm

SUMMARY:
Study GR40548 is a Phase III, randomized, multicenter, open-label (visual assessor [VA]-masked), active-comparator study designed to assess the efficacy, safety, and pharmacokinetics (PK) of 100mg/ml delivered via the Port Delivery System with ranibizumab (PDS) compared with ranibizumab intravitreal injections at 0.5 mg (10 mg/mL) in participants with neovascular age-related macular degeneration (nAMD).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥50 years, at time of signing Informed Consent Form
* Initial diagnosis of exudative neovascular age-related macular degeneration (nAMD) within 9 months prior to the screening visit
* Previous treatment with at least three anti-vascular endothelial growth factor (anti-VEGF) intravitreal injections for nAMD per standard of care within 6 months prior to the screening visit
* Demonstrated response to prior anti-VEGF intravitreal treatment since diagnosis
* Best-corrected visual acuity (BCVA) of 34 letters or better

Exclusion Criteria:

* Subfoveal fibrosis or subfoveal atrophy in study eye
* Subretinal hemorrhage that involves the center of the fovea in study eye
* History of vitrectomy surgery, submacular surgery, or other surgical intervention for AMD in study eye
* Prior treatment with Visudyne®, external-beam radiation therapy, or transpupillary thermotherapy in study eye
* Previous intraocular device implantation in study eye
* Previous laser (any type) used for AMD treatment in study eye
* Treatment with anti-VEGF agents other than ranibizumab within 1 month prior to the randomization visit in either eye
* Prior participation in a clinical trial involving anti-VEGF drugs within 6 months prior to the randomization visit, other than ranibizumab in either eye
* CNV due to other causes, such as ocular histoplasmosis, trauma, or pathologic myopia in either eye
* Uncontrolled blood pressure
* History of stroke within the last 3 months prior to informed consent
* Uncontrolled atrial fibrillation within 3 months of informed consent
* History of myocardial infarction within the last 3 months prior to informed consent
* History of other disease, metabolic dysfunction, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of ranibizumab or placement of the Implant and that might affect interpretation of the results of the study or renders the participant at high risk of treatment complications in the opinion of the investigator
* Current systemic treatment for a confirmed active systemic infection
* Chronic use of oral corticosteroids
* Active cancer within 12 months of randomization
* Previous participation in any non-ocular (systemic) disease studies of investigational drugs within 1 month preceding the informed consent (excluding vitamins and minerals)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 415 (Actual)
Dates: Start 2018-09-12 (Actual); Primary Completion 2020-05-22 (Actual); Study Completion 2021-06-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (77):
- United States (77):
  - Barnet Dulaney Perkins Eye Center, Mesa, Arizona
  - Associated Retina Consultants, Phoenix, Arizona
  - Arizona Retina and Vitreous Consultants, Phoenix, Arizona
  - Retinal Consultants of Arizona, Phoenix, Arizona
  - California Retina Consultants, Bakersfield, California
  - Retina-Vitreous Associates Medical Group, Beverly Hills, California
  - The Retina Partners, Encino, California
  - Jules Stein Eye Institute/ UCLA, Los Angeles, California
  - N CA Retina Vitreous Assoc, Mountain View, California
  - Retina Consultants, San Diego, Poway, California
  - Retinal Consultants Med Group, Sacramento, California
  - West Coast Retina Medical Group, San Francisco, California
  - UCSF; Ophthalmology, San Francisco, California
  - Orange County Retina Med Group, Santa Ana, California
  - California Retina Consultants, Santa Barbara, California
  - Bay Area Retina Associates, Walnut Creek, California
  - Southwest Retina Consultants, Durango, Colorado
  - Eye Center of Northern CO, Fort Collins, Colorado
  - Colorado Retina Associates, PC, Lakewood, Colorado
  - Retina Group of New England, Waterford, Connecticut
  - National Ophthalmic Research Institute, Fort Myers, Florida
  - Florida Eye Associates, Melbourne, Florida
  - Retina Care Specialists, Palm Beach Gardens, Florida
  - Retina Specialty Institute, Pensacola, Florida
  - Fort Lauderdale Eye Institute, Plantation, Florida
  - Retina Vitreous Assoc of FL, St. Petersburg, Florida
  - Southern Vitreoretinal Assoc, Tallahassee, Florida
  - Retina Associates of Florida, LLC, Tampa, Florida
  - Southeast Retina Center, Augusta, Georgia
  - Georgia Retina PC, Marietta, Georgia
  - Illinois Retina Associates, Joliet, Illinois
  - University Retina and Macula Associates, PC, Lemont, Illinois
  - Wolfe Eye Clinic, West Des Moines, Iowa
  - Retina Associates, Lenexa, Kansas
  - Retina Associates of Kentucky, Lexington, Kentucky
  - Paducah Retinal Center, Paducah, Kentucky
  - Maine Eye Center, Portland, Maine
  - The Retina Care Center, Baltimore, Maryland
  - Johns Hopkins Med; Wilmer Eye Inst, Baltimore, Maryland
  - Retina Group of Washington, Chevy Chase, Maryland
  - Retina Specialists, Towson, Maryland
  - Ophthalmic Consultants of Boston, Boston, Massachusetts
  - Vitreo-Retinal Associates, PC, Worcester, Massachusetts
  - Associated Retinal Consultants, Grand Rapids, Michigan
  - Foundation for Vision Research, Grand Rapids, Michigan
  - VitreoRetinal Surgery, PLLC.; DBA Retina Consultants of Minnesota, Edina, Minnesota
  - Midwest Vision Research Foundation, Chesterfield, Missouri
  - The Retina Institute - Chesterfield, Chesterfield, Missouri
  - Sierra Eye Associates, Reno, Nevada
  - Envision Ocular, LLC, Bloomfield, New Jersey
  - Mid Atlantic Retina - Wills Eye Hospital, Cherry Hill, New Jersey
  - NJ Retina Teaneck Clinic, Toms River, New Jersey
  - Long Is. Vitreoretinal Consult, Great Neck, New York
  - Retina Vit Surgeons/Central NY, Liverpool, New York
  - Vitreous-Retina-Macula, New York, New York
  - Ophthalmic Consultants of Long Island, Rockville Centre, New York
  - Char Eye Ear &Throat Assoc, Charlotte, North Carolina
  - Cincinnati Eye Institute, Cincinnati, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - OSU Eye Physicians & Surgeons, Columbus, Ohio
  - Retina Vitreous Center, Edmond, Oklahoma
  - Retina Northwest, Portland, Oregon
  - Palmetto Retina Center, Florence, South Carolina
  - Charles Retina Institute, Memphis, Tennessee
  - Tennessee Retina PC, Nashville, Tennessee
  - Texas Retina Associates, Arlington, Texas
  - Austin Retina Associates, Austin, Texas
  - Austin Clinical Research LLC, Austin, Texas
  - Retina Consultants of Texas, Bellaire, Texas
  - Texas Retina Associates, Fort Worth, Texas
  - Med Center Ophthalmology Assoc, San Antonio, Texas
  - Retina Associates of Utah, Salt Lake City, Utah
  - Rocky Mountain Retina, Salt Lake City, Utah
  - Wagner Macula & Retina Center, Norfolk, Virginia
  - Retina Institute of Virginia, Richmond, Virginia
  - Retina Center Northwest, Silverdale, Washington
  - Spokane Eye Clinical Research, Spokane, Washington

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.clinicalstudydatarequest.com). Further details on Roche's criteria for eligible studies are available here (https://clinicalstudydatarequest.com/Study-Sponsors/Study-Sponsors-Roche.aspx). For further details on Roche's Global Policy on Sharing of Clinical Study Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

REFERENCES:
- [Derived] Sheth VS, Holekamp NM, Khanani AM, Rachitskaya A, Blotner S, Gune S, Heinrich D, Maass KF, Chakravarthy U. Retinal Fluid and Thickness Fluctuations in Archway Trial for Port Delivery System with Ranibizumab versus Monthly Ranibizumab Injections. Ophthalmol Retina. 2025 Apr;9(4):330-342. doi: 10.1016/j.oret.2024.10.015. Epub 2024 Oct 22. PMID 39447871
- [Derived] Campochiaro PA, Eichenbaum D, Chang MA, Clark WL, Graff JM, Le Pogam S, Cavichini Cordeiro M, Gune S, Rabena M, Singh N, Lin S, Callaway N. Interim Results of the Phase III Portal Extension Trial of the Port Delivery System with Ranibizumab in Neovascular Age-Related Macular Degeneration. Ophthalmol Retina. 2025 Feb;9(2):144-155. doi: 10.1016/j.oret.2024.05.021. Epub 2024 Aug 30. PMID 39209113
- [Derived] Eichenbaum DA, Freeman WR, Chang MA, Brooks L, Chaudhry N, Dadgostar H, McCannel CA, Michels M, Mittra RA, Wolfe JD, Beindl VC, Jaycock P, Bobbala A, Gune S, Spicer G, Callaway N. Endophthalmitis in Eyes Treated with the Port Delivery System with Ranibizumab: Summary of Cases during Clinical Trial Development. Ophthalmol Retina. 2025 Feb;9(2):127-143. doi: 10.1016/j.oret.2024.08.005. Epub 2024 Aug 16. PMID 39154860
- [Derived] Nielsen JS, Chang A, Holekamp NM, Cavichini-Cordeiro M, Lin SL, Heinrich D, Maass KF, Menezes A, Singh N, Pieramici DJ. Supplemental Intravitreal Ranibizumab Injections in Eyes Treated with the Port Delivery System with Ranibizumab in the Archway Trial. Ophthalmol Retina. 2024 Dec;8(12):1127-1139. doi: 10.1016/j.oret.2024.06.012. Epub 2024 Jun 22. PMID 38914294
- [Derived] Chang MA, Kapre A, Kaufman D, Kardatzke DR, Rabena M, Patel S, Bobbala A, Gune S, Fung A, Wallenstein G. Patient Preference and Treatment Satisfaction With a Port Delivery System for Ranibizumab vs Intravitreal Injections in Patients With Neovascular Age-Related Macular Degeneration: A Randomized Clinical Trial. JAMA Ophthalmol. 2022 Aug 1;140(8):771-778. doi: 10.1001/jamaophthalmol.2022.1091. PMID 35708706
- [Derived] Awh CC, Barteselli G, Makadia S, Chang RT, Stewart JM, Wieland MR, Brassard R, Callaway NF, Gune S, Heatherton P, Malhotra V, Willis JR, Pieramici DJ. Management of Key Ocular Adverse Events in Patients Implanted with the Port Delivery System with Ranibizumab. Ophthalmol Retina. 2022 Nov;6(11):1028-1043. doi: 10.1016/j.oret.2022.05.011. Epub 2022 May 16. PMID 35589078
- [Derived] Heimann F, Barteselli G, Brand A, Dingeldey A, Godard L, Hochstetter H, Schneider M, Rothkegel A, Wagner C, Horvath J, Ranade S. A custom virtual reality training solution for ophthalmologic surgical clinical trials. Adv Simul (Lond). 2021 Apr 16;6(1):12. doi: 10.1186/s41077-021-00167-z. PMID 33863399

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PDS Implant Arm | Intravitreal Arm
Started | 248 | 167
Completed | 234 | 154
Not Completed | 14 | 13
Not completed — Adverse Event | 1 | 1
Not completed — Death | 8 | 4
Not completed — Lost to Follow-up | 3 | 0
Not completed — Non-Compliance With Study Drug | 1 | 0
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 1 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PDS Implant Arm | Intravitreal Arm | Total
Number analyzed (Participants) | 248 | 167 | 415
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 26 | 17 | 43
  >=65 years | 222 | 150 | 372
Age, Continuous [Mean (Standard Deviation); unit: Years] | 75.2 (8.11) | 74.8 (7.63) | 75.0 (7.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 145 | 100 | 245
  Male | 103 | 67 | 170
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 8 | 15
  Not Hispanic or Latino | 240 | 159 | 399
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 3
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 240 | 161 | 401
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Best-Corrected Visual Acuity (BCVA) Score at the Average of Week 36 and Week 40, as Assessed Using the ETDRS Visual Acuity Chart at a Starting Distance of 4 Meters
Description: The primary efficacy endpoint is the change in BCVA score from baseline averaged over Weeks 36 and 40 with BCVA assessed using the ETDRS chart at a starting distance of 4 meters. ETDRS = Early Treatment Diabetic Retinopathy Study.
  The primary objective is to determine the NI and equivalence between the two treatment groups, as measured by the primary efficacy endpoint with a NI margin of 4.5 letters and equivalence margins of ± 4.5 letters.
  A vision score of 20/20 vision is considered normal. A score of 20/200 is considered being legally blind.
Time Frame: Baseline, and the average of Week 36 and Week 40
Measure: Mean (95.03% Confidence Interval); unit: letters
Arm/Group | PDS Implant Arm | Intravitreal Arm
Number analyzed (Participants) | 248 | 167
letters | 0.2 [-0.7 to 1.1] | 0.5 [-0.6 to 1.6]

2. Secondary Outcome: Change From Baseline in BCVA Score Averaged Over Week 60 and Week 64
Time Frame: Baseline, Week60, Week 64
Population: Efficacy Population comprising all patients who are randomized and receive the study treatment, with patients grouped according to treatment actually received
Measure: Mean (95.03% Confidence Interval); unit: letters
Arm/Group | PDS Implant Arm | Intravitreal Arm
Number analyzed (Participants) | 248 | 167
letters | -0.4 [-1.5 to 0.7] | -0.8 [-2.2 to 0.6]

3. Secondary Outcome: Change From Baseline in BCVA Score Over Time
Time Frame: Baseline up to Week 96
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | PDS Implant Arm | Intravitreal Arm
Number analyzed (Participants) | 248 | 167
letters
  Week 4: number analyzed (Participants) | 246 | 165
  Week 4 | -4.3 (0.47) | -0.4 (0.58)
  Week 8: number analyzed (Participants) | 247 | 163
  Week 8 | -1.7 (0.41) | 0.1 (0.51)
  Week 12: number analyzed (Participants) | 244 | 161
  Week 12 | -0.4 (0.39) | 0.6 (0.48)
  Week 16: number analyzed (Participants) | 244 | 163
  Week 16 | -0.6 (0.41) | 0.2 (0.5)
  Week 20: number analyzed (Participants) | 242 | 163
  Week 20 | -0.3 (0.42) | 0.1 (0.52)
  Week 24: number analyzed (Participants) | 245 | 163
  Week 24 | -0.6 (0.47) | 0.8 (0.57)
  Week 28: number analyzed (Participants) | 243 | 162
  Week 28 | -0.1 (0.47) | 0.5 (0.57)
  Week 32: number analyzed (Participants) | 241 | 161
  Week 32 | 0.2 (0.49) | 0.9 (0.60)
  Week 36: number analyzed (Participants) | 242 | 160
  Week 36 | 0.2 (0.47) | 0.3 (0.58)
  Week 40: number analyzed (Participants) | 240 | 161
  Week 40 | 0.2 (0.51) | 0.7 (0.63)
  Week 44: number analyzed (Participants) | 234 | 157
  Week 44 | -0.1 (0.53) | 0.6 (0.65)
  Week 48: number analyzed (Participants) | 237 | 154
  Week 48 | 0.0 (0.53) | -0.2 (0.65)
  Week 52: number analyzed (Participants) | 209 | 144
  Week 52 | 0.1 (0.54) | -0.8 (0.67)
  Week 56: number analyzed (Participants) | 203 | 150
  Week 56 | 0.1 (0.56) | -0.5 (0.67)
  Week 60: number analyzed (Participants) | 209 | 154
  Week 60 | -0.5 (0.58) | -0.8 (0.71)
  Week 64: number analyzed (Participants) | 224 | 152
  Week 64 | -0.3 (0.59) | -0.7 (0.72)
  Week 68: number analyzed (Participants) | 230 | 153
  Week 68 | -0.5 (0.64) | -0.3 (0.79)
  Week 72: number analyzed (Participants) | 242 | 153
  Week 72 | -0.3 (0.64) | 0.1 (0.79)
  Week 76: number analyzed (Participants) | 224 | 149
  Week 76 | -1.0 (0.68) | 0.2 (0.83)
  Week 80: number analyzed (Participants) | 232 | 154
  Week 80 | -0.7 (0.64) | -0.2 (0.79)
  Week 84: number analyzed (Participants) | 225 | 153
  Week 84 | -0.8 (0.62) | 0.3 (0.77)
  Week 88: number analyzed (Participants) | 227 | 152
  Week 88 | -1.3 (0.62) | 0.0 (0.76)
  Week 92: number analyzed (Participants) | 218 | 148
  Week 92 | -0.9 (0.63) | -1.0 (0.78)
  Week 96: number analyzed (Participants) | 225 | 151
  Week 96 | -1.1 (0.68) | -1.3 (0.84)

4. Secondary Outcome: Percentage of Participants With BCVA Score of 38 Letters (20/200 Approximate Snellen Equivalent) or Worse at the Average Over Week 36 and Week 40
Time Frame: Baseline, and the average of Week 36 and Week 40
Population: Adult patients with nAMD diagnosed within 9 months and receiving at least 4 anti-VEGF intravitreal injections (with the last injection being ranibizumab), responsive to prior anti-VEGF treatment
Measure: Number (95.03% Confidence Interval); unit: Percentage of participants
Arm/Group | PDS Implant Arm | Intravitreal Arm
Number analyzed (Participants) | 248 | 167
Percentage of participants | 1.2 [0.0 to 2.6] | 1.8 [0.0 to 3.9]

5. Secondary Outcome: Percentage of Participants With BCVA Score of 38 Letters (20/200 Approximate Snellen Equivalent) or Worse Over Time
Time Frame: Baseline up to Week 96
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | PDS Implant Arm | Intravitreal Arm
Number analyzed (Participants) | 248 | 167
Percentage of Participants | 2.7 | 5.3

6. Secondary Outcome: Percentage of Participants With BCVA Score of 69 Letters (20/40 Approximate Snellen Equivalent) or Better at the Average Over Week 36 and Week 40
Time Frame: Baseline, and the average of Week 36 and Week 40
Population: as for outcome 4
Measure: Number (95.03% Confidence Interval); unit: Percentage of participants
Arm/Group | PDS Implant Arm | Intravitreal Arm
Number analyzed (Participants) | 248 | 167
Percentage of participants | 80.7 [76.9 to 84.5] | 82.1 [77.5 to 86.7]

7. Secondary Outcome: Percentage of Participants With BCVA Score of 69 Letters (20/40 Approximate Snellen Equivalent) or Better Over Time
Time Frame: Baseline up to Week 96
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | PDS Implant Arm | Intravitreal Arm
Number analyzed (Participants) | 248 | 167
Percentage of participants | 75.6 | 78.1

8. Secondary Outcome: Percentage of Participants Who Lose <10 or <5 Letters in BCVA Score From Baseline to the Average Over Week 36 and Week 40
Time Frame: Baseline, and the average of Week 36 and Week 40
Population: as for outcome 4
Measure: Number (95.03% Confidence Interval); unit: Percentage of participants
Arm/Group | PDS Implant Arm | Intravitreal Arm
Number analyzed (Participants) | 248 | 167
Percentage of participants
  Loss of Visual Function <10 letters | 95.1 [92.4 to 97.8] | 95.1 [91.8 to 98.4]
  Loss of Visual Function <5 letters | 85.0 [80.5 to 89.4] | 88.3 [83.4 to 93.3]

9. Secondary Outcome: Percentage of Participants Who Lose <10 or <5 Letters in BCVA Score From Baseline Over Time
Time Frame: Baseline up to Week 96
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | PDS Implant Arm | Intravitreal Arm
Number analyzed (Participants) | 248 | 167
Percentage of participants
  <10 letters | 88.9 | 84.1
  < 5 letters | 75.1 | 73.5

10. Secondary Outcome: Percentage of Participants Who Gain ≥0 Letters in BCVA Score From Baseline to the Average Over Week 36 and Week 40
Time Frame: Baseline up to Week 40
Population: as for outcome 4
Measure: Number (95.03% Confidence Interval); unit: Percentage of participants
Arm/Group | PDS Implant Arm | Intravitreal Arm
Number analyzed (Participants) | 248 | 167
Percentage of participants | 57.8 [51.8 to 63.7] | 58.9 [51.4 to 66.4]

11. Secondary Outcome: Percentage of Participants Who Gain ≥0 Letters in BCVA Score From Baseline Over Time
Time Frame: Baseline up to Week 96
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | PDS Implant Arm | Intravitreal Arm
Number analyzed (Participants) | 248 | 167
Percentage of Participants | 52.4 | 55.6

12. Secondary Outcome: Change From Baseline in Center Point Thickness (CPT) at Week 36
Time Frame: Baseline to Week 36
Population: Adult patients with nAMD diagnosed within 9 months and receiving at least 4 anti-VEGF intravitreal injections (with the last injection being ranibizumab), responsive to prior anti-VEGF treatment. 14 participants (7 participants in each arm) discontinued before Week 36 or the CPT value was missing (or not able to be measured on image) for the week 36 visit.
Measure: Mean (Standard Deviation); unit: microns
Arm/Group | PDS Implant Arm | Intravitreal Arm
Number analyzed (Participants) | 248 | 167
microns
  Baseline Value | 176.9 (3.48) | 177.4 (3.84)
  Week 36: number analyzed (Participants) | 241 | 160
  Week 36 | 5.4 (2.91) | 2.6 (3.56)

13. Secondary Outcome: Change From Baseline in CPT Over Time
Time Frame: Baseline up to Week 96
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: microns
Arm/Group | PDS Implant Arm | Intravitreal Arm
Number analyzed (Participants) | 248 | 167
microns
  Baseline Value: number analyzed (Participants) | 248 | 165
  Baseline Value | 176.9 (3.48) | 177.4 (3.84)
  Week 4: number analyzed (Participants) | 245 | 164
  Week 4 | 0.2 (2.05) | 2.1 (2.51)
  Week 8: number analyzed (Participants) | 247 | 162
  Week 8 | 0.3 (2.17) | 3.0 (2.66)
  Week 12: number analyzed (Participants) | 244 | 161
  Week 12 | 5.3 (2.87) | 0.3 (3.52)
  Week 16: number analyzed (Participants) | 244 | 163
  Week 16 | 6.0 (3.45) | 7.3 (4.23)
  Week 20: number analyzed (Participants) | 243 | 162
  Week 20 | 6.5 (2.7) | 1.3 (3.31)
  Week 24: number analyzed (Participants) | 243 | 163
  Week 24 | 6.7 (2.5) | -0.8 (3.06)
  Week 28: number analyzed (Participants) | 241 | 162
  Week 28 | -0.4 (2.5) | 1.6 (3.07)
  Week 32: number analyzed (Participants) | 239 | 162
  Week 32 | 4.5 (2.69) | 2.3 (3.29)
  Week 36: number analyzed (Participants) | 241 | 160
  Week 36 | 5.4 (2.91) | 2.7 (3.56)
  Week 40: number analyzed (Participants) | 238 | 161
  Week 40 | 9.0 (3.37) | 5.1 (4.13)
  Week 44: number analyzed (Participants) | 232 | 158
  Week 44 | 7.3 (3.13) | 3.4 (3.84)
  Week 48: number analyzed (Participants) | 237 | 153
  Week 48 | 8.9 (3.55) | 6.4 (4.36)
  Week 52: number analyzed (Participants) | 209 | 142
  Week 52 | 3.2 (3.43) | 6.6 (4.2)
  Week 56: number analyzed (Participants) | 201 | 151
  Week 56 | 2.7 (3.36) | 3.3 (4.10)
  Week 60: number analyzed (Participants) | 209 | 153
  Week 60 | 3.9 (3.39) | 2.5 (4.12)
  Week 64: number analyzed (Participants) | 224 | 152
  Week 64 | 5.5 (3.54) | 3.6 (4.34)
  Week 68: number analyzed (Participants) | 228 | 153
  Week 68 | 8.4 (3.48) | 2.1 (4.27)
  Week 72: number analyzed (Participants) | 238 | 152
  Week 72 | 8.1 (3.35) | 0.9 (4.14)
  Week 76: number analyzed (Participants) | 221 | 150
  Week 76 | 3.4 (3.61) | 0.1 (4.44)
  Week 80: number analyzed (Participants) | 230 | 153
  Week 80 | 6.1 (3.56) | -2.7 (4.38)
  Week 84: number analyzed (Participants) | 224 | 154
  Week 84 | 8.4 (3.87) | -2.0 (4.76)
  Week 88: number analyzed (Participants) | 225 | 151
  Week 88 | 9.8 (3.88) | -0.6 (4.77)
  Week 92: number analyzed (Participants) | 217 | 147
  Week 92 | 10.3 (3.57) | -1.3 (4.39)
  Week 96: number analyzed (Participants) | 222 | 151
  Week 96 | 9.9 (3.64) | -1.3 (4.48)

14. Secondary Outcome: Percentage of Participants in the PDS Implant Arm Who Undergo Supplemental Treatment With Intravitreal Ranibizumab 0.5 mg Before the First, Second, Third, and Fourth Fixed Refill-Exchange Intervals
Time Frame: Day 1 to Week 24, Week 25 to Week 48, Week 49 to Week 72, Week73 to Week 96
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | PDS Implant Arm
Number analyzed (Participants) | 246
Participants
  Day 1 to Week 24: Need for supplemental treatment | 4
  Day 1 to Week 24: No need for supplemental treatment | 242
  Week 25 to Week 48: number analyzed (Participants) | 241
  Week 25 to Week 48: Need for supplemental treatment | 13
  Week 25 to Week 48: No need for supplemental treatment | 228
  Week 49 to Week 72: number analyzed (Participants) | 231
  Week 49 to Week 72: Need for supplemental treatment | 12
  Week 49 to Week 72: No need for supplemental treatment | 219
  Week 73 to Week 96: number analyzed (Participants) | 225
  Week 73 to Week 96: Need for supplemental treatment | 12
  Week 73 to Week 96: No need for supplemental treatment | 213

15. Secondary Outcome: Percentage of Participants in the PDS Implant Arm Who Undergo a Supplemental Treatment That Requires Subsequent Additional Supplemental Treatments During the Study
Time Frame: Week 16 to Week 92
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | PDS Implant Arm
Number analyzed (Participants) | 246
Percentage of Participants
  2 supplemental treatments | 4.1
  3 supplemental treatments | 0.8
  5 supplemental treatments | 0.4

16. Secondary Outcome: Percentage of Participants With Ocular and Systemic (Non-Ocular) AEs
Time Frame: Randomization to Week 96
Population: Safety Population comprising all patients who receive the study treatment, with patients grouped according to treatment actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | PDS Implant Arm | Intravitreal Arm
Number analyzed (Participants) | 248 | 167
Participants
  Ocular Events: Study Eye | 242 | 87
  Ocular Events: Fellow Eye | 124 | 65
  Non-Ocular Events | 213 | 121

17. Secondary Outcome: Percentage of Participants With Adverse Events of Special Interest
Description: Percentage of Participants with Adverse Events of Special Interest
Time Frame: Randomization to Week 96
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | PDS Implant Arm | Intravitreal Arm
Number analyzed (Participants) | 248 | 167
Participants
  Adverse Events of Special Interest in Study Eye | 64 | 18
  Adverse Events of Special Interest in Fellow Eye | 21 | 6
  Non-Ocular Adverse Events of Special Interest | 0 | 0

18. Secondary Outcome: Observed Serum Ranibizumab Concentrations at Specified Timepoints
Time Frame: Randomization to Week 96
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PDS Implant Arm | Intravitreal Arm
Number analyzed (Participants) | 39 | 46
ng/mL
  Randomization: number analyzed (Participants) | 39 | 45
  Randomization | 0.125 (115) | 0.117 (78.5)
  Week 24 prerefill-exchange: number analyzed (Participants) | 36 | 44
  Week 24 prerefill-exchange | 0.397 (71.1) | 0.0592 (180)
  Week 28: number analyzed (Participants) | 28 | 35
  Week 28 | 0.564 (40.7) | 0.0581 (178)
  Week 48 prerefill-exchange: number analyzed (Participants) | 28 | 39
  Week 48 prerefill-exchange | 0.289 (90.6) | 0.0594 (146)
  Week 52: number analyzed (Participants) | 19 | 35
  Week 52 | 0.499 (41.7) | 0.0531 (123)
  Week 72 prerefill-exchange: number analyzed (Participants) | 29 | 30
  Week 72 prerefill-exchange | 0.257 (73.7) | 0.0376 (152)
  Week 76: number analyzed (Participants) | 19 | 32
  Week 76 | 0.291 (247) | 0.0500 (127)
  Week 96: number analyzed (Participants) | 33 | 41
  Week 96 | 0.191 (154) | 0.0680 (157)

19. Secondary Outcome: Estimated PK Parameter Values AUC0-6M
Description: AUC0-6M = Area Under the Concentration-Time Curve From 0 to 6 Months
Time Frame: Randomization to Week 96
Population: PK Population excluding patients receiving intravitreal injections of ranibizumab in the study eye post PDS implant (including supplemental treatment), patients with fellow eye ranibizumab or bevacizumab treatment, or prior bevacizumab treatment in either eye.
Measure: Mean (Standard Deviation); unit: day.ng/mL
Arm/Group | PDS Implant Arm
Number analyzed (Participants) | 33
day.ng/mL | 59.42 (21.11)

20. Secondary Outcome: Estimated PK Parameter Value t1/2 After PDS Implant Insertion
Description: Apparent terminal half-life
Time Frame: Randomization to Week 96
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: day
Arm/Group | PDS Implant Arm
Number analyzed (Participants) | 7
day | 442.29 (276.92)

21. Secondary Outcome: Estimated PK Parameter Value Cmin
Description: Cmin = Minimum Serum Concentration
Time Frame: Randomization to Week 96
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PDS Implant Arm
Number analyzed (Participants) | 33
ng/mL | 0.31 (0.08)

22. Secondary Outcome: Estimated PK Parameter Value Cmax
Description: Cmax = Maximum Serum Concentration
Time Frame: Randomization to Week 96
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PDS Implant Arm
Number analyzed (Participants) | 33
ng/mL | 0.47 (0.16)

23. Secondary Outcome: Baseline Prevalence and Incidence of Treatment-Emergent ADA
Time Frame: Randomization to Week 96
Population: The Biomarker Analysis Population consists of patients who are in the Safety Population and have sufficient data to enable assessment of potential changes in biomarkers in response to treatment during the conduct of this study. The analysis will group patients according to treatment actually received
Measure: Number; unit: Participants
Arm/Group | PDS Implant Arm | Intravitreal Arm
Number analyzed (Participants) | 248 | 167
Participants
  Patients with a positive sample at time of entry into the study: number analyzed (Participants) | 243 | 162
  Patients with a positive sample at time of entry into the study | 5 | 8
  Patients with no positive samples at time of entry into the study: number analyzed (Participants) | 243 | 162
  Patients with no positive samples at time of entry into the study | 238 | 154
  Post-baseline Patients Positive for ADA: number analyzed (Participants) | 247 | 165
  Post-baseline Patients Positive for ADA | 38 | 21
  Treatment-induced ADA: number analyzed (Participants) | 247 | 165
  Treatment-induced ADA | 33 | 15
  Treatment-enhanced ADA: number analyzed (Participants) | 247 | 165
  Treatment-enhanced ADA | 0 | 2
  Treatment unaffected or reduced: number analyzed (Participants) | 247 | 165
  Treatment unaffected or reduced | 5 | 6
  Patients negative for ADA at all times in the study: number analyzed (Participants) | 247 | 165
  Patients negative for ADA at all times in the study | 209 | 144

ADVERSE EVENTS:
Time Frame: Baseline up to 2 years
Arm/Group | Intravitreal Arm | PDS Implant Arm
All-Cause Mortality (participants affected / at risk) | 5/167 | 8/248
Serious Adverse Events (participants affected / at risk) | 39/167 | 78/248
Other Adverse Events (participants affected / at risk) | 58/167 | 225/248
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intravitreal Arm (N=167) | PDS Implant Arm (N=248)
Vitreous haemorrhage (Eye disorders) | 1 (1) | 2 (2)
Conjunctival erosion (Eye disorders) | 0 (0) | 3 (4)
Retinal tear (Eye disorders) | 1 (1) | 1 (1)
Visual acuity reduced (Eye disorders) | 0 (0) | 1 (4)
Cataract cortical (Eye disorders) | 0 (0) | 1 (1)
Conjunctival bleb (Eye disorders) | 0 (0) | 1 (1)
Corneal disorder (Eye disorders) | 0 (0) | 1 (1)
Retinal pigment epithelial tear (Eye disorders) | 0 (0) | 1 (1)
Rhegmatogenous retinal detachment (Eye disorders) | 0 (0) | 2 (3)
Choroidal detachment (Eye disorders) | 0 (0) | 1 (1)
Necrotising retinitis (Eye disorders) | 0 (0) | 1 (1)
Visual impairment (Eye disorders) | 0 (0) | 1 (1)
Endophthalmitis (Infections and infestations) | 1 (1) | 4 (5)
Conjunctival retraction (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 7 (7)
Sepsis (Infections and infestations) | 2 (2) | 3 (3)
Urinary tract infection (Infections and infestations) | 1 (1) | 6 (6)
Diverticulitis (Infections and infestations) | 0 (0) | 2 (2)
Cellulitis (Infections and infestations) | 2 (2) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 3 (3)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 2 (2)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 3 (3)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 4 (4)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (4)
Syncope (Nervous system disorders) | 3 (3) | 0 (0)
Disturbance in attention (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Parkinson's disease (Nervous system disorders) | 0 (0) | 1 (1)
Temporal lobe epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Acetabulum fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatic carcinoma stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Penile squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Small intestine adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma of pharynx (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Lactic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 2 (2)
Renal embolism (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal infarct (Renal and urinary disorders) | 0 (0) | 1 (1)
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Aortic stenosis (Vascular disorders) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Prostatomegaly (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1)
Aortic valve incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Retinal artery occlusion (Eye disorders) | 0 (0) | 1 (1)
Retinal haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Scleral thinning (Eye disorders) | 0 (0) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mesenteric vein thrombosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 3 (3) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1)
Mucosal inflammation (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Gallbladder rupture (Hepatobiliary disorders) | 1 (1) | 0 (0)
Arthritis infective (Infections and infestations) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Kidney infection (Infections and infestations) | 1 (2) | 0 (0)
Metapneumovirus pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1)
Post procedural infection (Infections and infestations) | 0 (0) | 1 (1)
Septic arthritis staphylococcal (Infections and infestations) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 2 (2)
Device dislocation (Product Issues) | 0 (0) | 3 (3)
Hip arthroplasty (Surgical and medical procedures) | 1 (1) | 0 (0)
Aortic aneurysm (Vascular disorders) | 0 (0) | 1 (1)
Arteriosclerosis (Vascular disorders) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intravitreal Arm (N=167) | PDS Implant Arm (N=248)
Conjunctival haemorrhage (Eye disorders) | 12 (14) | 178 (193)
Conjunctival hyperaemia (Eye disorders) | 3 (4) | 66 (71)
Iritis (Eye disorders) | 1 (1) | 50 (55)
Eye pain (Eye disorders) | 8 (8) | 25 (28)
Vitreous floaters (Eye disorders) | 4 (4) | 23 (24)
Vitreous detachment (Eye disorders) | 8 (11) | 17 (19)
Punctate keratitis (Eye disorders) | 4 (6) | 17 (25)
Vitreous haemorrhage (Eye disorders) | 3 (4) | 13 (14)
Neovascular age-related macular degeneration (Eye disorders) | 15 (15) | 20 (20)
Foreign body sensation in eyes (Eye disorders) | 2 (2) | 18 (20)
Hypotony of eye (Eye disorders) | 0 (0) | 15 (15)
Conjunctival bleb (Eye disorders) | 0 (0) | 16 (16)
Nasopharyngitis (Infections and infestations) | 14 (15) | 13 (14)
Headache (Nervous system disorders) | 4 (4) | 14 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2021-02-02): https://cdn.clinicaltrials.gov/large-docs/34/NCT03677934/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-09): https://cdn.clinicaltrials.gov/large-docs/34/NCT03677934/SAP_001.pdf